CLINICAL TRIAL: NCT00214942
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of ORAVESCENT Fentanyl Citrate for Management of Breakthrough Pain in Opioid-Tolerant Patients With Chronic Low Back Pain
Brief Title: Study to Evaluate the Efficacy and Safety of ORAVESCENT Fentanyl Citrate for Management of Breakthrough Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: C25608/3042/BP/US
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Low Back Pain

INTERVENTIONS:
Drug: ORAVESCENT Fentanyl Citrate

SUMMARY:
A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of ORAVESCENT Fentanyl Citrate for Management of Breakthrough Pain in Opioid-Tolerant Patients with Chronic Low Back Pain

ELIGIBILITY:
Inclusion Criteria:

Patients are included in the study if all of the following criteria are met:

* The patient is willing to provide written informed consent to participate in this study.
* The patient is 18 through 80 years of age.
* Women must be surgically sterile, 2 years postmenopausal, or, if of childbearing potential, using a medically accepted method of birth control (ie, barrier method with spermicide, steroidal contraceptive [oral, transdermal, implanted, or injected contraceptives must be used in conjunction with a barrier method], or intrauterine device [IUD]) and agree to continued use of this method for the duration of this study.
* The patient has a diagnosis of chronic low back pain, resulting in functional disability of at least 3 months duration and is associated with any of the following: osteoarthritis, degenerative disc disease, or spondylolisthesis. Patients with other low back pain etiologies may qualify for the study with permission from the Cephalon medical monitor or designee.
* The patient is currently using 1 of the following: at least 60 mg/day or oral morphine/day, or at least 25 mcg transdermal fentanyl/hour, or at least 30 mcg oxycodone/day, as a stable dose of around-the-clock (ATC) therapy for at least the previous 7 days before enrollment into the study.
* The patient reports an average pain intensity score, over the prior 24 hours, of less than 7 (0=no pain through 10=worst pain) for their chronic low back pain.
* The patient experiences, on average, 1 to 4 BTP episodes (defined as temporary flares of severe or excruciating pain) per day while taking ATC opioid therapy, and on average, the duration of each BTP episode is less than 4 hours.
* The patient currently uses opioid therapy for alleviation of BTP episodes, occuring at the location of the chronic pain, and achieves at least partial relief.
* The patient is able to effectively self-administer the study drug.

Exclusion Criteria:

Patients are excluded from participating in this study if 1 or more of the following criteria are met:

* The patient has uncontrolled or rapidly escalating pain as determined by the investigator (ie, the ATC therapy may be expected to change between the first and last treatments with study drug), or has pain uncontrolled by therapy that could adversely impact the safety of the patient or that could be compromised by treatment with study drug.
* The patient has known or suspected hypersensitivities, allergies, or other contraindications to any ingredient in the study drug.
* The patient has a recent history (within 5 years) or current evidence of alcohol or other substance abuse.
* The patient has cardiopulmonary disease that would, in the opinion of the investigator, significantly increase the risk of treatment with potent synthetic opioids.
* The patient has medical psychiatric disease that, in the opinion of the investigator, would compromise collected data.
* The patient is expected to have surgery during the study and it is anticipated that the surgery will alleviate the patient's pain.
* The patient has had therapy before study drug treatment that, in the opinion of the investigator, could alter pain or response to pain medication.
* The patient is pregnant or lactating.
* The patient has participated in a previous study with ORAVESCENT fentanyl.
* The patient has participated in a study involving an investigational drug in the previous 30 days.
* The patient has received a monoamine oxidase inhibitor (MAOI) within 14 days before the first treatment with study drug.
* The patient has any other medical condition or is receiving concomitant medication/therapy (eg, regional nerve block) that would, in the opinion of the investigator, compromise the patient's safety or compliance with the study protocol, or compromise collected data.
* The patient is involved in active litigation in regard to their chronic pain.
* The patient has a positive urine drug screen (UDS) for a medication not prescribed by their physician or no reasonable explanation can be provided to the Cephalon medical monitor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-09; Primary Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Clopton Clinic, Jonesboro, Arkansas
  - Vertex Clinical Research, Inc., Bakersfield, California
  - San Diego Arthritis Medical, San Diego, California
  - Clinical Research of W Florida, Clearwater, Florida
  - Florida Institute of Medical R, Jacksonville, Florida
  - Clinical Pharmacology Services, Tampa, Florida
  - Gold Coast Research, Weston, Florida
  - Center for Prospective Outcome, Marietta, Georgia
  - Georgia Medical Research, Marietta, Georgia
  - American Medical Research, Chicago, Illinois
  - American Medical Research, Oak Brook, Illinois
  - American Medical Research, Valparaiso, Indiana
  - Iowa Pain Management Clinic, P, Des Moines, Iowa
  - Mid America Physiatrists, PA, Overland Park, Kansas
  - Best Clinical Trial, Inc., New Orleans, Louisiana
  - PharmQuest, Greensboro, North Carolina
  - Northwest Clinical Research, Bellevue, Washington